CLINICAL TRIAL: NCT00844038
Title: Stevens-Johnson Syndrome Associated With Antimicrobial
Brief Title: Stevens-Johnson Syndrome Antimicrobial
Status: Completed | Type: Observational
Sponsor: University of Pernambuco (Other)
Responsible Party: Stevens-Johnson syndrome associated with antimicrobial, University of Pernambuco
Other Study IDs: SSJ1; 558187121279
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Last update posted 2009-02-13 (Estimated); Status verified 2009-02

CONDITIONS: Stevens-Johnson Syndrome
Keywords: Steven-Johnson syndrome; erythema multiform; autoimmune disease
MeSH Terms: conditions — Stevens-Johnson Syndrome; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Sick

SUMMARY:
Steven-Johnson's syndrome, or great multiform erythema, appears as a systemic disturbance, with skin involvement and mucous membranes, related to several factors, such as, viral or bacterial infections and mainly the administration of medicines, in general painkillers and antibiotics. The objective of this work is report the emergence of ulcerative vesicle -bubble chronic disease in areas of lips, gum, tongue and genital mucous membrane in a 26 year-old patient, leucoderma and masculine gender, in treatment of breathing infection with sulfametoxazol-trimetropima, having been diagnosed as syndrome of Steven-Johnson.

DETAILED DESCRIPTION:
Among the serious medicaments reactions, there are as great representative the Mucocutaneous Disorders immunological mediated. Steven-Johnson's syndrome, or great multiform erythema, appears as a systemic disturbance, with skin involvement and mucous membranes, related to several factors, such as, viral or bacterial infections and mainly the administration of medicines, in general painkillers and antibiotics. The objective of this work is report the emergence of ulcerative vesicle -bubble chronic disease in areas of lips, gum, tongue and genital mucous membrane in a 26 year-old patient, leucoderma and masculine gender, in treatment of breathing infection with sulfametoxazol-trimetropima, having been diagnosed as syndrome of Steven-Johnson.

ELIGIBILITY:
Inclusion Criteria:

* Stevens-Johnson syndrome associated with antimicrobial

Exclusion Criteria:

* Not sick

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: 1
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-08; Primary Completion 2008-08 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edwaldo Dr Dourado, Doctor, Principal Investigator — University of Pernambuco
Locations (1):
- University of Pernambuco, Recife, Pernambuco, Brazil

REFERENCES:
- [Result] Vanfleteren I, Van Gysel D, De Brandt C. Stevens-Johnson syndrome: a diagnostic challenge in the absence of skin lesions. Pediatr Dermatol. 2003 Jan-Feb;20(1):52-6. doi: 10.1046/j.1525-1470.2003.03012.x. PMID 12558848